CLINICAL TRIAL: NCT03441581
Title: 3030-401-002: An Open-Label Pilot Study of Eluxadoline in Participants With Irritable Bowel Syndrome With Diarrhea (IBS-D) Who Have Evidence of Bile Acid Malabsorption (BAM)
Brief Title: Eluxadoline Bile Acid Malabsorption (BAM) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3030-401-002
Record Dates: First submitted 2018-01-19; First posted 2018-02-22 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS-D; BAM
MeSH Terms: interventions — eluxadoline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eluxadoline 100 mg with BAM (Experimental): IBS-D participants with evidence of Bile Acid Malabsorption (BAM) treated with eluxadoline 100 mg oral tablets twice daily (BID) with food for 4 weeks.
  Interventions: Drug: Eluxadoline
- Eluxadoline 100 mg without BAM (Experimental): IBS-D participants without evidence of BAM treated with eluxadoline 100 mg oral tablets BID with food for 4 weeks.
  Interventions: Drug: Eluxadoline

INTERVENTIONS:
Drug: Eluxadoline — Eluxadoline 100 mg oral tablets BID with food.

SUMMARY:
This study will evaluate the possibility of a differential effect of eluxadoline on altered bowel function in Irritable Bowel Syndrome with Diarrhea (IBS-D) participants with and without evidence of Bile Acid Malabsorption (BAM).

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18 to 75 years inclusive with a diagnosis of IBS-D per Rome IV criteria.
* Participants with evidence of BAM must have a fasting serum 7a-hydroxy-4-cholesten-3-one (7αC4) level ≥ 52.5 ng/mL or total fecal bile acid (BA) > 2337 micromoles/48 hours (positive result) at screening or within 1 calendar year prior to screening.
* Participants without BAM must have a fasting serum 7αC4 level ≤ 47.1 ng/mL or total fecal BA < 2200 micromoles/48 hours (negative result) at screening or within 1 calendar year prior to screening.
* Has an average daily Bristol Stool Form Scale (BSFS) score ≥ 5.0 or ≥ 25% of diary entry days with a BSFS score of 6 or 7 during the 14 days prior to Day 1.
* Women of childbearing potential must use hormonal or double barrier contraception or maintain a monogamous relationship with a vasectomized male partner from the date of informed consent until 24 hours after final dose of study drug.
* Completed the electronic diary (eDiary) on ≥ 10 of the 14 days prior to Day 1.
* Has not used loperamide rescue medication on > 3 of the 14 days prior to Day 1.

Exclusion Criteria:

* Has a diagnosis of IBS with a subtype of irritable bowel syndrome with constipation (IBS-C), mixed IBS, or unsubtyped IBS per Rome IV criteria.
* Does not have a gallbladder.
* Has known or suspected biliary duct obstruction, or sphincter of Oddi disease or dysfunction. (Participants with a history of gallstones may be enrolled).
* Has a history of alcoholism, alcohol abuse or alcohol addiction, or drinks more than 3 alcoholic beverages per day.
* Has a history of pancreatitis; structural diseases of the pancreas, including known or suspected pancreatic duct obstruction.
* Has a history of mild, moderate, or severe hepatic impairment according to Child-Pugh classification. History or current diagnosis of inflammatory or immune-mediated gastrointestinal (GI) disorders.
* Has Celiac disease or a positive serological test for celiac disease.
* Has known lactose or fructose intolerance associated with diarrhea, abdominal pain or discomfort, that could confound assessments in the study.
* Women who are currently pregnant or nursing, or plan to become pregnant or nurse during the study.
* Has known allergies or hypersensitivity to opioids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Muslin, Study Director — Allergan
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included of all participants who received ≥ 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (6.07) | 40.2 (13.72) | 40.9 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Bristol Stool Form Scale (BSFS) Score Over 4 Weeks of Treatment Period
Description: Stool consistency was assessed using the BSFS where: 1=Separate hard lumps like nuts to 7=Watery. The score was recorded by the participant in an electronic diary (e-diary). The score for each day was averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: Modified Intent-to-Treat (mITT) Population included of all participants in Enrolled Population with ≥ 1 postbaseline assessment for BSFS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 5.89 (0.639) | 5.34 (0.777)
  Change From Baseline at Week 4 | -1.25 (0.914) | -1.09 (0.902)

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is an AE that occurs or worsens after receiving investigational study drug.
Time Frame: Baseline (Day 1) to Week 4
Population: Safety Population included of all participants who received ≥ 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
percentage of participants | 91.7 | 58.3

3. Primary Outcome: Number of Participants Who Experienced Potentially Clinically Significant Change in Laboratory Tests
Description: Laboratory tests included tests of Clinical Chemistry, Hematology, and Urinalysis. The investigator determined if the result was potentially clinically significant.
Time Frame: Baseline (Day 1) to Week 4
Population: Safety Population included of all participants who received ≥ 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
Participants | 0 | 2

4. Primary Outcome: Number of Participants Who Experienced Potentially Clinically Significant Change in Vital Signs
Description: Vital signs assessments included: pulse, respiratory rate, and blood pressure (systolic and diastolic). The investigator determined if the result was potentially clinically significant.
Time Frame: Baseline (Day 1) to Week 4
Population: Safety Population included of all participants who received ≥ 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1

5. Primary Outcome: Number of Participants Who Experienced Clinically Significant Change From Baseline in General Physical Condition as Measured Through General Physical Exam
Description: General Physical Examination consisted of a full review of body systems excluding pelvic and rectal exams. The investigator determined if the result was clinically significant.
Time Frame: Baseline (Day 1) to Week 4
Population: Safety Population included of all participants who received ≥ 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

6. Secondary Outcome: Change From Baseline in the 4-week Average of Daily Bowel Movement Frequency During the Treatment Period
Description: Bowel movements were recorded by the participant in an electronic diary (e-diary). The number of bowel movements per day was averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS.
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
bowel movements per day
  Baseline | 4.18 (2.792) | 2.86 (1.071)
  Change from Baseline at Week 4 | -1.48 (1.509) | -0.79 (0.420)

7. Secondary Outcome: Change From Baseline in the 4-week Average of Daily Worst Abdominal Pain Scores During the Treatment Period
Description: The participant recorded their worst abdominal pain score in the past 24 hours each day in an e-diary where: 0=no pain to 10=worst imaginable pain. The score each day was averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 1.77 (1.510) | 3.13 (1.755)
  Change from Baseline at Week 4 | -0.12 (0.769) | -1.28 (1.004)

8. Secondary Outcome: Change From Baseline in the 4-week Average of Daily Bloating Scores During the Treatment Period
Description: The participant recorded their bloating score in the past 24 hours each day in an e-diary where: 0=no bloating to 10=worst imaginable bloating. The score each day was averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 2.31 (2.291) | 4.07 (2.496)
  Change from Baseline at Week 4 | -0.47 (1.572) | -1.46 (1.297)

9. Secondary Outcome: Change From Baseline in the 4-week Average Number of Daily Urgent Bowel Movements During the Treatment Period
Description: The participant recorded the number of urgent bowel movements in the past 24 hours each day in an e-diary. The number of urgent bowel movements per day was averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS.
Measure: Mean (Standard Deviation); unit: urgent bowel movements per day
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
urgent bowel movements per day
  Baseline | 1.67 (1.179) | 1.22 (0.652)
  Change from Baseline at Week 4 | -0.52 (0.736) | -0.80 (0.651)

10. Secondary Outcome: Percentage of Participants With Any Fecal Incontinence During the Treatment Period
Description: The participant recorded the number of fecal incontinences in the past 24 hours each day in an e-diary. Fecal incontinence is the inability to control the passage of gas or stools. The number of fecal incontinences per day was averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
percentage of participants | 33.3 | 33.3

11. Secondary Outcome: Change From Baseline in Irritable Bowel Syndrome Quality of Life (IBS-QOL) Total Score at the End of the Treatment Period
Description: IBS-QOL is composed of 34 items about how the symptoms of IBS are impacting the participant's life scored on a 1 to 5 scale, where lower item scores indicate greater quality of life. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0 to 100-point scale (0=worst; 100=better) for ease of interpretation. A positive change from Baseline indicates improved quality of life.
Time Frame: Baseline (Day1) to End of Treatment (Up to Week 4)
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 75.1 (14.43) | 71.4 (13.42)
  Change from Baseline at Week 4 | 8.8 (11.70) | 13.2 (10.63)

12. Secondary Outcome: Change From Baseline in Fasting Serum 7α-hydroxy-4-cholesten-3-one (7αC4) Levels at the End of the Treatment Period
Description: Participants fasted for at least 8 hours prior to the test. Fasting serum 7αC4 level was measured at Baseline and End of Treatment to determine whether any changes occurred following treatment with eluxadoline. The negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to End of Treatment (Up to Week 4)
Population: mITT Population included of all participants in enrolled population with ≥ 1 postbaseline assessment for BSFS. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
nanogram/milliliter (ng/mL)
  Baseline | 42.95 (27.259) | 30.58 (17.248)
  Change from Baseline at End of Treatment: number analyzed (Participants) | 10 | 12
  Change from Baseline at End of Treatment | -5.59 (32.841) | -8.78 (12.050)

13. Secondary Outcome: Cmax: Maximum Concentration for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: Pharmacokinetic (PK) population included all participants in the enrolled population and whose dry blood sample (DBS) was collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
ng/mL | 1.40 (1.34) | 0.91 (0.80)

14. Secondary Outcome: Cmin: Minimum Concentration for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: PK population included all participants in the enrolled population and whose DBS was collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
ng/mL | 0.39 (0.44) | 0.42 (0.59)

15. Secondary Outcome: AUC: Area Under the Concentration-time Curve During the Dosing Interval for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: PK population included all participants in the enrolled population and whose DBS was collected.
Measure: Mean (Standard Deviation); unit: nanogram* hour/milliliter (ng*h/mL)
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
nanogram* hour/milliliter (ng*h/mL) | 9.22 (8.46) | 7.75 (8.48)

16. Secondary Outcome: Tmax: Time to Cmax for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: PK population included all participants in the enrolled population and whose DBS was collected.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
hours (h) | 1.5 [1.0 to 2.5] | 2.0 [1.0 to 3.0]

17. Secondary Outcome: t1/2: Half-Life for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: PK population included all participants in the enrolled population and whose DBS was collected.
Measure: Median (Full Range); unit: h
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
h | 30.5 [24.7 to 58.1] | 35.2 [24.7 to 88.6]

18. Secondary Outcome: CL/F: Apparent Total Clearance of the Drug From Plasma After Oral Administration for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: PK population included all participants in the enrolled population and whose DBS was collected.
Measure: Mean (Standard Deviation); unit: liter/hour (L/h)
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
liter/hour (L/h) | 20236 (13280) | 21901 (11921)

19. Secondary Outcome: Vc/F: Apparent Volume of Distribution for Eluxadoline
Time Frame: Predose and at the intervals 1-2, 3-4 and 5-8 hours postdose at Week 2
Population: PK population included all participants in the enrolled population and whose DBS was collected.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
Number analyzed (Participants) | 12 | 12
L | 29432 (11000) | 39799 (10637)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Eluxadoline 100 mg With BAM | Eluxadoline 100 mg Without BAM
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline 100 mg With BAM (N=12) | Eluxadoline 100 mg Without BAM (N=12)
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Flatulence (Gastrointestinal disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03441581/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03441581/SAP_001.pdf